CLINICAL TRIAL: NCT03052803
Title: Comparison of Devices Evaluating Fractional Flow Reserve in Coronary Arteries : FRACTIONAL FLOW RESERVE - DEVICE STUDY (FFR-DS)
Brief Title: Comparison of Devices Evaluating Fractional Flow Reserve in Coronary Arteries
Acronym: FFR-DS
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Collaborators: Acist Medical Systems (Industry); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-145
Record Dates: First submitted 2017-02-10; First posted 2017-02-14 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2017-12

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Myocardial Ischemia
Keywords: coronary stenosis; fractional flow reserve
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Fractional flow reserve measure — Comparison of different devices measuring fractional flow reserve

SUMMARY:
The aim of the study is to compare different devices available to measure fractional flow reserve (FFR) in coronary arteries.

DETAILED DESCRIPTION:
The decision to perform a percutaneous coronary intervention (PCI) is usually based on angiographic results alone. Angiography can be used for the visual evaluation of the inner diameter of a vessel. Visual evaluation is limited by inter-individual variability.

Fractional flow reserve provides a functional evaluation, by measuring the pressure decline caused by a vessel narrowing.

The original studies validating the use of FFR were conducted with only one device (St-Jude Medical®). Recently, new FFR devices have been commercialized but have not yet been compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized at Caen University Hospital for coronary angiography
* Coronary stenosis needing FFR evaluation according to recommendations
* More than 18 years old
* Clinically stable
* De novo coronary stenosis
* Affiliated to social security
* Informed consent signed

Exclusion Criteria:

* Unstable patients defined by acute coronary syndrome < 7 days
* Contre-indication to adenosine administration (asthma, allergy, high grade atrio-ventricular bloc without pace maker)
* History of coronary artery bypass
* intra-stent restenosis
* Patient not capable of understanding the study
* Informed consent not signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutifs patients hospitalized for coronary angiography and presenting one or several coronary stenosis needing FFR evaluation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Simultaneous FFR measure SJM and ACIST | Immediately
  Correlation between simultaneous measures with St Jude medical FFR device and ACIST device
Simultaneous FFR measure Boston Scientific and ACIST | Immediately
  Correlation between simultaneous measures with BOSTON Scientific FFR device and ACIST device
Simultaneous FFR measure Boston Scientific and SJM | Immediately
  Correlation between simultaneous measures with BOSTON Scientific FFR device and St Jude Medical device

SECONDARY OUTCOMES:
FFR SJM or Boston alone versus simultaneous with ACIST | Immediately
  Correlation between SJM and Boston Scientific FFR measurements alone and simultaneous measure with ACIST
Clinical concordance | Immediately
  Concordance between FFR values >0.80 or <=0.80
Drift of the signal | immediately
  variation between the initial measure in the aorta (equalization) and final measure

CONTACTS AND LOCATIONS:
Locations (1):
- CAEN University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: No